CLINICAL TRIAL: NCT00674622
Title: Prolotherapy for the Treatment of Chronic Lateral Epicondylitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Ronald M. Glick, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R21AT003969-01A1 (NIH); 1R21AT003969-01A1 (NIH)
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Lateral Epicondylitis; Tennis Elbow
Keywords: Lateral epicondylitis; Tennis elbow; Prolotherapy
MeSH Terms: conditions — Tennis Elbow | interventions — Prolotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1-Prolotherapy (Experimental): Deep injection with 15% dextrose in lidocaine
  Interventions: Drug: Prolotherapy
- Group 2-Deep Saline/Lidocaine (Placebo Comparator): Deep injection with saline/lidocaine
  Interventions: Procedure: Placebo
- Group 3-Superficial Saline/lidocaine (Placebo Comparator): Superficial injection with saline/lidocaine
  Interventions: Procedure: Placebo

INTERVENTIONS:
Drug: Prolotherapy — Injection of 15% dextrose with lidocaine at the lateral epicondyle
  Arms: Group 1-Prolotherapy
Procedure: Placebo — Saline/lidocaine
  Arms: Group 2-Deep Saline/Lidocaine; Group 3-Superficial Saline/lidocaine

SUMMARY:
Lateral epicondylitis (LE), or tennis elbow, is a common and often disabling condition affecting young and middle-aged adults-most commonly manual workers and recreational athletes. It results in significant pain and disability, limiting work productivity and an individual's ability to participate in and enjoy recreational activities. Like many other chronic musculoskeletal conditions LE often shows an incomplete response to acute treatments, leading to chronic pain and disability. Prolotherapy (PrT) involves the injection of an irritant or proliferant solution into tendons, ligaments, and joints to treat chronic musculoskeletal pain. We will be conducting a 3-group randomized, blinded trial to determine the safety and efficacy of PrT injections in the treatment of chronic LE. Additionally, we will seek to determine to what extent any beneficial effect of PrT is derived from deep needle placement vs. a specific effect of the injectate. The specific aims for this study are: 1) to determine if PrT is a safe, well-tolerated, and effective treatment for individuals with chronic LE; and 2) to determine whether the deep needle placement alone is responsible for the therapeutic effect, independent of injectate. In order to accomplish these aims, we will measure indicators of pain and disability using self-rating scales, questionnaires and physical measures. Subjects will be stratified prior to randomization on two factors: 1) unilateral vs. bilateral LE; and 2) treatment with steroids within the prior 6 months. If effective, subjects receiving PrT will show greater reduction of pain and functional impairment compared with the other two groups. This research will guide future studies on prolotherapy by determining what may be the best control condition. Additionally, further studies may explore the mechanism responsible for any beneficial effect.

DETAILED DESCRIPTION:
Same

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-65, as younger individuals are more likely to have other developmental conditions and older individuals are more likely to have a significant arthritic component to their elbow pain;
2. Ability to speak, read, and write English;
3. Unilateral or bilateral lateral elbow pain associated with findings on exam consistent with LE and absence of other conditions that can mimic LE such as radial tunnel syndrome.
4. Functional impairment, due to the diagnosis of LE, with a Nirschl Pain Phase Scale (NPPS) rating of Phase 4 or higher.

Exclusion Criteria:

1. Other conditions that result in significant impairment in upper extremity function such as fibromyalgia, rotator cuff tendonitis, cervical radiculopathy, or carpal tunnel syndrome;
2. Prior surgery of the involved elbow;
3. Known allergy to lidocaine or dextrose;
4. Presence of an autoimmune condition such as rheumatoid arthritis, given that a possible immune mechanism is hypothesized for PrT.
5. Presence of known immune dysfunction, such as with HIV/AIDS, as it might raise the risk for development of infection from injections;
6. Ongoing treatment with systemic corticosteroids or immunosuppressant medications, as they may block a potential immune mechanism of the PrT and increase the risk for infection;
7. Active diagnosis of malignancy anywhere in the body, given potential of any concurrent immune dysfunction to impact on the response to PrT;
8. Treatment with any anticoagulant medication beyond 1 aspirin per day, given the potential to increase bleeding or bruising associated with injections;
9. Presence of a coagulopathy, given the potential to increase bleeding or bruising associated with injections;
10. Pregnancy-as there is no research documenting safety of PrT during pregnancy;
11. Medical necessity for taking ongoing nonsteroidal anti-inflammatory medication, beyond 1 aspirin per day for cardiac prevention, as this may diminish the effect of PrT;
12. Corticosteroid injection within the 6 weeks prior to entry into the study, as this may diminish the effect of the PrT.
13. Prior treatment with PrT for any condition, as this may impact on blinding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-09; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Glick, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Center for Integrative Medicine at UPMC Shadyside, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Presented at conference.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between 3/17/2008 to 3/15/2010. All patients were seen at the University of Pittsburgh Medical Center outpatient clinics.
Pre-assignment Details: 105 subjects completed informed consent.
  38 subjects were ineligible, based on absence of diagnosis of lateral epicondylitis, insufficient severity of symptoms, or presence of an exclusion.
  1 subject completed all assessments but declined participation and was not randomized.
Period: Overall Study
Arm/Group | Group 1-Prolotherapy | Group 2-Deep Saline/Lidocaine | Group 3-Superficial Saline/Lidocaine
Started | 22 | 22 | 22
Completed | 21 | 18 | 22
Not Completed | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1-Prolotherapy | Group 2-Deep Saline/Lidocaine | Group 3-Superficial Saline/Lidocaine | Total
Number analyzed (Participants) | 22 | 22 | 22 | 66
Age, Continuous [Mean (Full Range); unit: years] | 49 [32 to 64] | 50 [34 to 65] | 50 [39 to 63] | 49 [32 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 11 | 28
  Male | 15 | 12 | 11 | 38
Race/Ethnicity, Customized [Number; unit: participants]
  White | 18 | 22 | 22 | 62
  Black | 2 | 0 | 0 | 2
  Asian | 1 | 0 | 0 | 1
  Hispanic | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 22 | 66

OUTCOME MEASURES:

1. Primary Outcome: McGill Pain Questionnaire
Description: This is a pain severity rating. 15 adjectival descriptors of pain are scored on a 0-3 scale for a total score of 0-45 with a high score reflecting greater pain severity.
Time Frame: 6 weeks and 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1-Prolotherapy | Group 2-Deep Saline/Lidocaine | Group 3-Superficial Saline/Lidocaine
Number analyzed (Participants) | 22 | 22 | 22
units on a scale
  Baseline | 16.6 (9.0) | 15.7 (6.4) | 14.3 (6.2)
  End of Phase 1 | 8.2 (7.7) | 8.4 (6.0) | 6.0 (6.4)
  End of Phase 2 | 5.6 (5.5) | 3.7 (3.9) | 5.4 (4.8)

2. Secondary Outcome: QuickDASH
Description: The QuickDASH is an abbreviated form of the rating scale DASH or Disabilities of the Arm, Shoulder, & Hand. This is a self-report rating of function for individuals with problems of the upper extremity. The Institute for Work and Health, in collaboration with the American Academy of Orthopaedic Surgeons developed a self-report questionnaire "Disabilities of the Arm, Shoulder, & Hand". It is seen as a valid and reliable measure of upper extremity functional impairment, is in widespread use in the States and abroad, having been translated into multiple languages and has been used for studies on LE. 11 items are scored on this self-rating instrument on a 1-5 Likert scale with higher score reflecting greater disability. The scores are averaged and then converted to a 100 point scale (0-100), with higher score reflecting greater disability.
Time Frame: 6 weeks and 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1-Prolotherapy | Group 2-Deep Saline/Lidocaine | Group 3-Superficial Saline/Lidocaine
Number analyzed (Participants) | 22 | 22 | 22
units on a scale
  Baseline | 40.2 (16.2) | 39.7 (15.6) | 32.5 (16.0)
  End of Phase 1 | 18.5 (18.6) | 21.2 (17.3) | 16.7 (17.5)

3. Secondary Outcome: Grip Strength
Description: Maximal pain-free grip strength has been used as a physical correlate of disability associated with LE. Grip strength was obtained using a Jamar Dynamometer set in the 2nd position. 3 trials were recorded and the average pain-free grip strength was noted.
Time Frame: 6 weeks and 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Group 1-Prolotherapy | Group 2-Deep Saline/Lidocaine | Group 3-Superficial Saline/Lidocaine
Number analyzed (Participants) | 22 | 22 | 22
pounds
  Baseline | 52.18 (26.03) | 57.31 (34.96) | 60.89 (25.09)
  End of Phase 1 | 65.28 (20.89) | 67.87 (30.38) | 78.54 (27.07)
  End of Phase 2 | 66.87 (20.90) | 78.70 (30.76) | 82.17 (28.83)

4. Secondary Outcome: Nirschl Pain Phase Scale
Description: The Nirschl Pain Phase Scale (NPPS), which has been used to describe functional impairment related to tendinopathies such as lateral epicondylitis. This scale provides a global rating of impairment associated with sports and musculoskeletal injuries. A rating from 0-7 describes the phase of overuse injuries, with Phase 0 noting "No stiffness or soreness after activity" and Phase 7 corresponding with "Pain that also disrupts sleep consistently. Pain is aching in nature and intensifies with activity". It was used as an indication of severity for entry into the study and as the criterion for treatment response.
Time Frame: 6 and 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1-Prolotherapy | Group 2-Deep Saline/Lidocaine | Group 3-Superficial Saline/Lidocaine
Number analyzed (Participants) | 22 | 22 | 22
units on a scale
  Baseline | 5.18 (0.66) | 5.18 (0.85) | 5.23 (0.92)
  End of Phase 1 | 2.86 (1.96) | 3.17 (1.86) | 2.32 (1.39)
  End of Phase 2 | 2.10 (1.51) | 2.19 (0.91) | 2.09 (1.31)

5. Secondary Outcome: Pain Threshold on Dolorimetry
Description: Pressure pain threshold (PPT) has been noted to correlate with pain and disability associated with LE. PPT was determined by applying pressure with a digital algometer over the area of maximal tenderness corresponding with the common extensor tendon area. Only 1 determination was obtained as the 1st application of pressure can lower the pain threshold for subsequent testing.
Time Frame: 6 and 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Group 1-Prolotherapy | Group 2-Deep Saline/Lidocaine | Group 3-Superficial Saline/Lidocaine
Number analyzed (Participants) | 22 | 22 | 22
Pounds
  Baseline | 6.34 (2.71) | 6.37 (2.72) | 7.67 (2.85)
  End of Phase 1 | 8.26 (3.08) | 7.87 (3.75) | 9.81 (4.57)
  End of Phase 2 | 9.68 (3.05) | 10.13 (4.44) | 11.57 (5.45)

ADVERSE EVENTS:
Arm/Group | Group 1-Prolotherapy | Group 2-Deep Saline/Lidocaine | Group 3-Superficial Saline/Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes